CLINICAL TRIAL: NCT05870982
Title: Effects of Early vs. Late Time Restricted Eating vs. Daily Caloric Restriction on Weight Loss and Metabolic Outcomes in Adults With Obesity
Brief Title: Early vs. Late Time Restricted Eating vs. Daily Caloric Restriction
Acronym: Time2Eat
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 22-1829; R01DK132372 (NIH)
Record Dates: First submitted 2023-05-04; First posted 2023-05-23 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-12

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: randomized, parallel-arm clinical trial
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Early time restricted eating (Experimental): Participants will asked to follow early time restricted eating
  Interventions: Behavioral: Early TRE
- Late time restricted eating (Experimental): Participants will be asked to follow late time restricted eating
  Interventions: Behavioral: Late TRE
- Daily caloric restriction (Active Comparator): Participants will be instructed to follow daily caloric restriction
  Interventions: Behavioral: DCR

INTERVENTIONS:
Behavioral: Early TRE — Participants will be instructed to eat only during an 8-hour window starting 1-2 hours after waking.
  Arms: Early time restricted eating
Behavioral: Late TRE — Participants will be instructed to eat only during an 8-hour window starting 5-6 hours after waking.
  Arms: Late time restricted eating
Behavioral: DCR — Participants will be instructed to reduce caloric intake by 25%.
  Arms: Daily caloric restriction

SUMMARY:
The goal of this clinical trial is to learn about time restricted eating as a weight loss intervention in adults with obesity. The main questions it aims to answer are:

1. How does the timing of the eating window (early vs late time restricted eating) affect weight loss and changes in metabolic risk factors?
2. How does time restricted eating compare to standard of care (daily caloric restriction) for weight loss and changes in metabolic risk factors?

Participants will be randomly assigned to either early time restricted eating, late time restricted eating, or daily caloric restriction.

1. They will be asked to follow the assigned dietary strategy for 1 year and will receive a group-based program for instruction and support.
2. They will be asked at several times during the year to have their weight and body composition measured, provide blood samples, track their food, and wear monitors for physical activity and sleep.

DETAILED DESCRIPTION:
This is a 52-week randomized, parallel-arm clinical trial designed to assess the effects of early time restricted eating (E-TRE) vs late TRE (L-TRE) vs daily caloric restriction (DCR) within the context of a guidelines-based behavioral weight loss program. 162 adults (age 18-65) with obesity (BMI 27-45 kg/m2) will be recruited from the community and randomized 1:1:1 to E-TRE (eating within an 8-hour window starting 1-2 hours after waking), L-TRE (eating within an 8-hour window starting 5-6 hours after waking) or DCR (caloric restriction of 25% from baseline energy requirements). The primary outcome is change in body weight at 26 weeks. Secondary outcomes include body composition, insulin sensitivity, blood pressure, glucose variability, physical activity, and sleep.

ELIGIBILITY:
Inclusion Criteria:

* Adult males and females with a BMI of 27-45 kg/m2
* Age, 18-65 years old
* Passing medical and physical screening, and analysis of blood and urine screening samples
* Individuals who are not currently following an intermittent fasting or TRE dietary regimen (i.e., eating across less than a 10-hour period during the day).
* Own a smartphone
* Live or work within 45 minutes of the Anschutz Health & Wellness Center (exceptions may be made at the discretion of the Study PI on a case-by-case basis for highly motivated subjects)
* No plans to relocate within the next 12 months
* Capable and willing to give informed consent, understand exclusion criteria, and accept the randomized group assignment.
* Have a primary care physician (or are willing to establish care with a primary care physician prior to study enrollment) to address medical issues which may arise during screening or study procedures/interventions.

Exclusion Criteria:

* Pregnancy or lactation for women (women who are >6 months postpartum with no plans of becoming pregnant in the next year and who are not currently lactating can be included; oral contraceptives will be allowed if medication has been consistent for the prior 6 months)
* Weight loss >5kg in past 3 months for any reason except post-partum weight loss, weight gain >5kg in past 3 months requires assessment by PI to determine reason for weight gain and if it is appropriate for the subject to participate in the study
* Weight loss of >50 lbs in past 3 years for any reason except post-partum weight loss
* Presence or history of any metabolic or chronic health problems which would affect appetite, food intake, energy metabolism, or ability to optimally participate in the exercise component including: CVD, peripheral vascular disease, cerebrovascular disease, significant cardiac arrhythmias or cardiac valve disease, diabetes, uncontrolled hyper- or hypothyroidism, uncontrolled hypertension, cancer (within the last 5 years, except skin cancer or other cancers considered cured with excellent prognosis), HIV infection, seizure disorders, significant gastrointestinal disorders (described below), significant pulmonary disorders (described below), significant renal, musculoskeletal, neurologic, hematologic, or psychiatric disease.
* Significant gastrointestinal disorders including: chronic malabsorptive conditions, peptic ulcer disease, Crohn's disease, Ulcerative Colitis, chronic diarrhea, or active gallbladder disease.
* Significant pulmonary disorders including: chronic obstructive pulmonary disease (COPD), interstitial lung disease, cystic fibrosis, or uncontrolled asthma.
* Symptoms suggestive of CVD: chest pain, shortness of breath at rest or with mild exertion, syncope.
* Taking medications affecting weight or energy intake/energy expenditure in the last 6 months, including weight loss medications, antipsychotic drugs or other medications as determined by the study physician
* Having abnormal blood chemistry (eGFR<45mL/min, AST or ALT >3 times the upper limit of normal) or as deemed significant by the study physician
* LDL cholesterol >200 mg/dL
* Triglycerides > 500 mg/dL
* Being considered unsafe to participate as determined by the study physician
* Previous obesity treatment with surgery or weight loss device, except: (1) liposuction and/or abdominoplasty if performed > 1 year before screening, (2) lap banding if the band has been removed > 1 year before screening, (3) intragastric balloon if the balloon has been removed > 1 year before screening (4) duodenal-jejunal bypass sleeve, if the sleeve has been removed > 1 year before screening or 5) AspireAssist or other endoscopically placed weight loss device if the device has been removed > 1 year before screening.
* Being a smoker or having been a smoker in the 3 months prior to their screening visit
* Working night shifts
* Night eating syndrome (at least 25% of food intake is consumed after the evening meal and/or at least two episodes of nocturnal eating per week) as assessed with meal pattern assessment questionnaire
* History of clinically diagnosed eating disorders including anorexia nervosa, bulimia, binge eating disorder. Score >20 on the EATS-26, score of >27 on the BES, or pattern of response on the QEWP-5 suggestive of possible binge eating disorder or bulimia will require further assessment by the Study MD to determine if it is appropriate for the subject to participate in the study.
* Current alcohol or substance abuse (assessed with CAGE-AID questionnaire (48))
* Current severe depression or history of severe depression within the previous year, based on DSM-IV-TR criteria for Major Depressive Episode. Score > 18 on BDI will require further assessment by the Study MD to determine if it is appropriate for the subject to participate in the study.
* Individuals who are already following an intermittent fasting or TRE dietary regimen and individuals not willing to abstain from alcohol outside of prescribed eating windows will also be excluded.
* Currently participating in or planning to participate in any formal weight loss or physical activity programs or clinical trials
* Regular use of systemic steroids (other than oral contraceptive pills)
* Medication(s) that must be taken with food (PI discretion based on whether it would be feasible for the participant to take the medication with food in the afternoon or evening if assigned to L-TRE group)
* Currently participating in a weight loss program or research study or participation in a weight loss program or research study within 1 year prior to intervention start date.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2023-07-11 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Body weight (kg) | 0 to 52 weeks
  Body weight will be measured using a digital scale at baseline, weeks 14, 26 and 52. The primary outcome will be change in weight from baseline to 26 weeks.

SECONDARY OUTCOMES:
Fat mass | 0 to 52 weeks
  Fat mass will assessed using Dual-Energy X-Ray Absorptiometry (DXA) at baseline, weeks 14, 26 and 52
Lean mass | 0-52 weeks
  Lean mass will assessed using Dual-Energy X-Ray Absorptiometry (DXA) at baseline, weeks 14, 26 and 52
Blood pressure | 0-52 weeks
  Systolic and diastolic blood pressure will be measured at baseline and weeks 14, 26 and 52
HbA1c | 0-52 weeks
  HbA1c will be measured at baseline and weeks 14, 26 and 52
Insulin sensitivity | 0-52 weeks
  Insulin sensitivity measured with oral glucose tolerance test at baseline and weeks 14, 26 and 52
24-hour glucose levels | 0-52 weeks
  24-hr glucose levels measured with continuous glucose monitor at baseline and weeks 14, 26 and 52
Physical activity | 0-52 weeks
  Total steps measured with activPal device at baseline and weeks 14, 26 and 52
Total cholesterol concentration | 0-52 weeks
  Total cholesterol concentration will be measured at baseline and weeks 14, 26 and 52
Sleep duration | 0-52 weeks
  Sleep duration (minutes) will be measured with activPal device at baseline and weeks 0, 14 and 26
LDL cholesterol concentration | 0-52 weeks
  Low density lipoprotein (LDL) will be measured at baseline and weeks 14, 26 and 52
HDL cholesterol concentration | 0-52 weeks
  High density lipoprotein (HDL) cholesterol concentration will be measured at baseline and weeks 14, 26 and 52
Triglyceride concentration | 0-52 weeks
  Triglyceride concentration will be measured at baseline and weeks 14, 26 and 52

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado Anschutz Health and Wellness Center, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No